CLINICAL TRIAL: NCT02857049
Title: Effective Consumption of Oral Nutritional Supplements in Geriatrics: A Study Evaluating a Strategy Based on a Preliminary Degustation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013-03
Record Dates: First submitted 2016-07-27; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Malnutrition; Geriatric Patients
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

ARMS (1):
- Geriatric patients administered with ONS (Experimental): Oral nutritional supplements (ONS) degustation
  Interventions: Other: Oral nutritional supplements (ONS) degustation

INTERVENTIONS:
Other: Oral nutritional supplements (ONS) degustation

SUMMARY:
Malnutrition affects until 70% of the patients hospitalized in geriatric's units and constitutes an independent risk factor of morbidity and mortality. Malnutrition is also associated with increased length of stay and increased costs, and alters the quality of life. Oral nutritional supplements (ONS) play a key role in the prevention and treatment of malnutrition in older people. ONS are a simple way to offer in a small volume a nutritional supply with a high density of calorie and protein. The clinical efficiency of ONS is well demonstrated whether on nutritional parameters or on clinical outcomes. However, acceptability and consumption of these ONS are frequently suboptimal: in geriatrics, only 50% to 65% of the prescribed volumes of ONS are consumed. The reasons are multiple: anorexia, taste changes, monotony … also partly because patients dislike flavor, taste or texture. The respect of patients' preferences is essential to improve the therapeutic observance to ONS. Generally, ONS are delivered after the patient has told his preferences orally to the dietitian. To date, there is no study evaluating the effect of an alternative strategy based on a preliminary degustation of several products on the effective consumption of ONS in geriatrics.

The study is designed as prospective, randomized, controlled, open study to test this strategy in older undernourished people hospitalized in geriatrics who require prescription of ONS. This study will be performed among 220 older people hospitalized in two departments of geriatrics of the AP-HM (Assistance Publique - Hôpitaux de Marseille).

The main objective is to compare the therapeutic observance to ONS when products are delivered to older people according to the usual way (preferences announced orally and/or dietitian's choice) or according to an alternative strategy based on a preliminary degustation of several products varying for flavor and texture but always in respect of the medical prescription. The secondary objective is to compare the evolution of the nutritional status estimated by routinely used clinical and biological parameters, as well as the main clinical outcomes during the hospital stay. Lastly, the nutritional status of these patients will be reevaluated clinically 3 months after the hospital's discharge.

The hypothesis is that a strategy based on a preliminary degustation, leading to an informed choice, will significantly improve the acceptability and the effective consumption of ONS during the hospital stay, and will also impact positively the nutritional status at hospital's discharge and 3 months after. The validation of this hypothesis could allow recommending the generalization of preliminary degustation of ONS at the time of their prescription to optimize the therapeutic observance in undernourished older people.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 70 years, hospitalized in a geriatric service for a short stay
* Patient malnourished or at risk of malnutrition, justifying the medical prescription of ONS
* Patient agreeing to participate in the study and who signed the informed consent form

Exclusion Criteria:

* Patient particularly protected (adult and incapable person deprived of liberty)
* Patient with a disease making it impossible to administer oral feeding
* Patient for which it is impossible to gather enough reliable data interrogation (dementia, pre-dementia, lack of proficiency in the French language)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of the consumed quantity of ONS in weight percentage | 3 months
Assessment of the consumed quantity of ONS in weight percentage | 3 months after hospital's discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France